CLINICAL TRIAL: NCT00971269
Title: A Pilot Study of Intersphincteric Injection of NASHA/Dx Gel for Fecal Incontinence
Brief Title: Pilot Study of NASHA/Dx Gel for Fecal Incontinence
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Professor Wilhelm Graf, Dept of Surgery, Uppsala University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPN 2008/066
Record Dates: First submitted 2009-09-02; First posted 2009-09-03 (Estimated); Last update posted 2009-09-03 (Estimated); Status verified 2009-09

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Solesta (Nasha/Dx) — Gel (hyaluronic acid/dextranomer) for intersphincteric injection 4x2 ml and retreatment 4x2 ml after 4 weeks
  Other Names: Solesta

SUMMARY:
The study is an open, prospective, single-site study where 16 patients suffering from fecal incontinence will be included. Change in fecal incontinence episodes after intersphincteric injection of NASHA/Dx gel 4x2 ml and retreatment 4x2 ml after 4 weeks will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Fecal incontinence with at least 2 episodes/week
2. Symptom duration at least one year
3. Failed attempt of conservative therapy
4. Age 18-80
5. Written informed consent
6. Available for follow-up
7. Fully compliant with protocol

Exclusion Criteria:

1. Active inflammatory bowel disease
2. Total external sphincter defect at ultrasound and clinical examination
3. Bleeding diathesis or anticoagulant therapy
4. Rectal prolapse or intussusceptions
5. Present anal sepsis
6. Anorectal implants
7. Recent anorectal surgery (within 6 months)
8. Rectal anastomosis
9. Pregnancy, postpartum (one year) or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Change in fecal incontinence episodes | Follow up during a four week period and after 6 and 12 months

SECONDARY OUTCOMES:
Side effects related to treatment | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, University Hospital, 751 82 Uppsala, Sweden